NCT03868631

Official title: Muscle growth and development following a 12-week resistance training program in

men and women consuming soy and whey protein supplements.

Date: August 1, 2016

Statistical analyses

Some outcomes were transformed using log10 transformation (lean body mass, peak torque for leg extensions, visceral adipose tissue (VAT), and bone mineral density) or square root transformation (peak torque for leg flexions) to achieve normality. Between-arm differences at baseline were compared using independent t-tests. Age was non-normal and thus baseline differences were assessed using a Mann Whitney U Test. Multilevel models for change (MLM) were used to determine differences between arms over time for study outcomes. Age, sex, and number of sessions missed were included as covariates. Study outcomes tested were total body mass; lean body mass; fat mass; body fat percent; bone mineral density; leg extension peak torque; leg flexion peak torque; and total kcal, carbohydrate, protein, and fat consumed. Time (categorical) and time by study arm interaction effects were examined. Time was also included as a random effect for the intercept to improve model fit and to account for individual differences in change over time. Lean body mass and subcutaneous adipose tissue models failed to converge when including the number of sessions missed as a covariate (fixed effect); therefore, this variable was removed from the model for these two outcomes. Data shown in Tables 3-5

reflect multi-level modeling with all participants who started the training (N=31 whey, 30 soy). All

analyses were conducted using IBM SPSS Statistics version 23.